CLINICAL TRIAL: NCT05134519
Title: Phase II Clinical Study to Evaluate the Efficacy and Safety of Recombinant Humanized Anti-HER2 Monoclonal Antibody-MMAE Coupling Agent (RC48-ADC) for Neoadjuvant Treatment of Breast Cancer With Positive HER2 Expression (Seraph)
Brief Title: RC48 for Neoadjuvant Chemotherapy of HER2 Positive Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XJLL-KY20212136
Record Dates: First submitted 2021-09-23; First posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-09

CONDITIONS: Breast Cancer; HER2-positive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RC48 for neadjuvant chemotherapy (Experimental): RC48-ADC: 2.0 mg/kg, IV drip, Q2W
  Interventions: Drug: Recombinant humanized anti-HER2 monoclonal antibody-MMAE coupling agent (RC48-ADC)

INTERVENTIONS:
Drug: Recombinant humanized anti-HER2 monoclonal antibody-MMAE coupling agent (RC48-ADC) — Regimen: RC48-ADC: 2.0 mg/kg, intravenous drip, once every 2 weeks,4-6 cycles
  Other Names: RC48

SUMMARY:
This is a single-arm exploratory study to explore the effect of RC48 in HER2-positive neoadjuvant therapy and evaluate the non-inferiority of RC48 by comparing the latest reported data of T-DM1 in neoadjuvant therapy.

DETAILED DESCRIPTION:
A single-arm exploratory study was conducted in 20 patients with HER2-positive breast cancer to explore the effect of RC48 in HER2-positive neoadjuvant therapy (treatment regimen: RC482.0 mg/kg, intravenous drip, once every 2 weeks). After 4-6 cycles, surgery was performed to evaluate the effect of neoadjuvant chemotherapy. The latest reported data of T-DM1 in neoadjuvant therapy were compared to evaluate the non-inferiority of RC48.

ELIGIBILITY:
Inclusion Criteria:

1. Enrolled were ≥ 18 years of age and < 80 years of age
2. Female or male breast cancer
3. Patients with early or locally advanced breast cancer who are HER2-positive, have a tumor larger than 2 cm and/or have lymph node metastasis: HER2-positive is defined as 3 + by immunohistochemistry, or 2 + by immunohistochemistry, with a positive FISH test.
4. Left ventricular score ≥ 55%
5. ECOGPS score 0 or 1
6. Able to understand the test requirements, willing and able to comply with the test and follow-up procedures
7. Adequate organ function

Exclusion Criteria:

1. cardiac, hepatic, renal, or psychiatric disease history
2. History of other malignancy within the last 5 years, with the exception of adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-11-26 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate (pCR) | At the end of Cycle 1 (each cycle is 14 days)
  absence of invasive carcinoma in the breast and axillary lymph nodes, while residual ductal carcinoma in situ was accepted (ypT0orTisypN0).

SECONDARY OUTCOMES:
adverse effects | during the period of neadjuvant chemotherapy
  Serious adverse effect occur within neoadjuvant chemotherapy

IPD SHARING:
Plan to Share IPD: No